CLINICAL TRIAL: NCT05895500
Title: An Investigator-Initiated Phase 2a, Open-Label Study to Evaluate the Safety and Efficacy of CGRP Antagonists in Patients With Dry Eye Disease and Asthenopia
Brief Title: Evaluate the Safety and Efficacy of Calcitonin Gene-Related Peptide (CGRP) Antagonists in Patients With Dry Eye Disease and Asthenopia
Status: Completed | Type: Observational
Sponsor: Nvision Laser Eye Centers (Industry)
Responsible Party: Sponsor
Other Study IDs: PPM_IIS_101
Record Dates: First submitted 2023-05-19; First posted 2023-06-08 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Dry Eye; Asthenopia
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia | interventions — Injections; Syringes; Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 56 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tablet: Tablets (50mg/tablet), oral
  Interventions: Drug: Tablet (50mg/tablet), oral
- Injection: Injection for SC administration (120mg/syringe)
  Interventions: Drug: Injection for SC administration (120mg/syringe)

INTERVENTIONS:
Drug: Injection for SC administration (120mg/syringe) — Injection
  Groups: Injection
Drug: Tablet (50mg/tablet), oral — Tablet
  Groups: Tablet

SUMMARY:
Safety and Efficacy of Medications for Migraine in Patients with Dry Eye Disease or Asthenopia

DETAILED DESCRIPTION:
An Investigator-Initiated Phase 2a, Open-Label Study to Evaluate the Safety and Efficacy of Medications for Migraine in Patients with Dry Eye Disease or Asthenopia

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the key components of the study as described in the written ICF, and willing and able to provide written informed consent.
2. Male or female ≥ 18 years of age.
3. Clinical diagnosis of:

   * Dry eye disease with episodes of eye discomfort in at least 4 of the previous 28 days during medical history assessment at Screening Visit, and have intensity >40 mm on a VAS scale at Screening (Day -28) visit OR
   * Asthenopia with episodes of eye discomfort in at least 4 of previous 28 days during medical assessment at Screening Visit and have intensity > 40 mm on a VAS scale at Screening (Day -28) visit. The cause of asthenopia should be recorded.
4. Willing and able to comply with the study requirements including prohibited concomitant medication restrictions.
5. Agree not to participate in another interventional study while on treatment.
6. If female, is surgically sterile or 2 years postmenopausal. Women of childbearing potential may be enrolled if a urine pregnancy test is negative at Screening and at Baseline Visits. Women of childbearing potential and men with partners who are of childbearing potential must agree to use highly effective methods of contraception from Screening throughout the study. Contraception use must continue for 90 days after the last administration of the study drug. Examples of acceptable methods of contraception which must be used together are described in Section 14.
7. If male, agrees to use a medically accepted highly effective method of contraception, agrees to use this method for 90 days after last administration of the study drug, and agrees to not donate sperm for 90 days after last administration of the study drug
8. Agree not to change lifestyle significantly during this study (Day -28 to Day 28).

Exclusion Criteria:

1. Active ocular infection or ocular inflammatory disease other than dry eye disease
2. Presence of anterior membrane dystrophy or history of clinically significant recurrent erosion syndrome.
3. Significant hematologic, endocrine, cardiovascular, cerebrovascular, pulmonary, renal, hepatic, gastrointestinal, or neurologic disease.
4. Prior radial keratotomy at any time or prior laser refractive surgery within the past 12 months of Screening Visit.
5. Unable to discontinue any over the counter (OTC), herbal, or systemic administration (including transdermal applications) of opioids or treatments for neuropathic pain (e.g., gabapentin or pregabalin, tetrahydrocannabinol) during the study on Days -28 to +28.
6. Seated blood pressure > 140 mmHg (systolic) or > 90 mmHg (diastolic).
7. History (within the past 30 days) or currently taking strong or moderate cytochrome P450 3A4 (CYP3A4) inhibitors (e.g., itraconazole, ketoconazole, fluconazole; erythromycin, clarithromycin, telithromycin; diltiazem, verapamil; aprepitant, cyclosporine, grapefruit juice, and HIV protease inhibitors), strong or moderate CYP3A4 inducers (e.g., barbiturates, primidone, mitotane, enzalutamide, efavirenz, apalutamide, carbamazepine, phenytoin, rifampin, , and St. John's wort), inhibitors of the BCRP (breast cancer resistance protein) transporter (e.g., curcumin and eltrombopag), and/or P-gp inhibitors (e.g., clarithromycin, quinidine, and cyclosporine), or drugs with narrow therapeutic margins (e.g., digoxin, warfarin). For a more complete list see FDA https://www.fda.gov/drugs/drug-interactions-labeling/drug- development and-drug-interactions-table-substrates-inhibitors-and-inducers#table5-2 (August 24, 2022).
8. Pregnant or plans to become pregnant and/or patients who are breastfeeding or plan to breastfeed during the study.
9. Current malignancy or a history of malignancy (within the past 5 years), except non metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
10. Significant liver disease, defined as having elevated aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels greater than 1.5 times the upper value of the normal range of the laboratory OR total bilirubin greater than 1.5 mg/dL (except for patients with a diagnosis of Gilbert's disease) OR serum albumin less than 2.8 g/dL at Screening Visit.
11. History of any other acute or chronic medical condition or pre-planned medical/surgical procedure that, in the opinion of the Investigator, would compromise the safety of the patient or the integrity of study results.
12. History of acute hepatitis within 6 months of Screening Visit or chronic hepatitis (including nonalcoholic steatohepatitis) or a positive result on anti-hepatitis A immunoglobulin M (IgM) antibody, hepatitis B surface antigen, or anti-hepatitis C antibody testing at Screening Visit.
13. Concurrent participation in another interventional study or treatment with an investigational drug up to 30 days or 5 half-lives (depending on medication) prior to Screening Visit.
14. Any form of substance abuse, psychiatric disorder, or a condition that, in the opinion of the Investigator, could invalidate communication with the Investigator during the study.
15. Positive test result for drugs of abuse at Screening Visit.
16. Unable to have a stable routine at home and workplace during the study.
17. The Principal Investigator reserves the right to declare a patient ineligible based on medical evidence that indicates the patient is unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from the clinical database that have previous symptoms and/or chief complaints of dry eye syndrome and asthenopia.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Tablet group | 28 Days
  Improvement in Symptoms: Number of days that a participant feels improvement in subjective symptoms of eye discomfort due to DED or asthenopia after oral administration of tablets over the 28-day Treatment Period (Days 1 to 28) compared to the 28-day Pretreatment Period (Day -28 to Day -1).
Injection group | 28 Days
  Improvement in Symptoms: Number of subjective symptom-free days due to DED or asthenopia over the 28-day Treatment Period (Days 1 to 28), following a single injection compared to the Pretreatment Period (Day -28 to Day -1).

SECONDARY OUTCOMES:
All Treatment Groups | 28 Days
  Change from baseline in visual analog scale (VAS) scores related to eye discomfort to EoS. A decrease in VAS scores while under the treatment will show the efficacy of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ahn, Principal Investigator — Employee for the Platform
Locations (1):
- NVision-EWEI-Torrance, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No